CLINICAL TRIAL: NCT02729415
Title: Point-of-Care Adipose-derived Cells for Hair Growth
Acronym: ASVF-2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201600420; ASVF-2016 (Other: Protocol)
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Androgenetic Alopecia
Keywords: Hair Diseases; Alopecia
MeSH Terms: conditions — Alopecia; Hair Diseases | interventions — Injections; Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal Vascular Fraction Cells (SVF Cells) (Experimental): The participants will undergo a standard tumescent liposuction to harvest adipose tissue. The adipose tissue will then be processed for obtain the Stromal Vascular Fraction Cells (SVF Cells) for a single injection for the treatment of androgenetic alopecia. Before the procedure, hair measurements will be performed in the 2cm x 2cm site for density (number of hairs per square centimeter) and thickness (mm) of the hair to compare to the measurements after the procedure at pre-procedure, 6 weeks, 3 months and 6 months.
  Interventions: Procedure: Stromal Vascular Fraction Cells (SVF Cells) Injection; Procedure: Liposuction; Other: Hair Measurements

INTERVENTIONS:
Procedure: Stromal Vascular Fraction Cells (SVF Cells) Injection — The procedure involves the injection of stromal vascular fraction cells (SVF Cells) into the scalp. The injection will be performed once in the middle of two perpendicular sides of a 2 x 2 cm area.
  Other Names: SVF Cells
Procedure: Liposuction — Tissue collection involving the micro-harvest of subcutaneous adipose tissue to harvest the stromal vascular fraction cells (SVF Cells).
  Other Names: Collection of adipose tissue
Other: Hair Measurements — Hair measurements will be performed using a computerized handheld USB camera at baseline, 6 weeks, and months 3 and 6 after treatment.

SUMMARY:
Androgenetic alopecia (AGA) is the most common form of hair loss and affects 50% and 23% of Caucasian men and women, respectively, over the age of 50. The percentage of men and women affected over the age of 70 increases to 80% and 60% of Caucasian men and women, respectively. Although alopecia is considered a minor dermatologic condition, it is seen as a serious condition with major life consequences by those with alopecia and has been associated with increased incidence of myocardial infarction, hypertension and hypercholesterolaemia. Androgenetic alopecia is associated with feelings of anxiety, depression and various personality disorders among men and women due to physical appearance. Depression, anxiety, aggressiveness, impaired quality of life and social inadequacy have been documented. The presence of alopecia in women is particularly stressful.

ADSCs (Adipose Derived Stromal Cells), also called Stromal Vascular Fraction (SVF) cells, include regenerative cell populations derived from adipose tissue and thus are potentially important to multiple disease processes and therapeutic applications for the repair and regeneration of acute and chronically damaged tissues. It has been postulated that SVF cells may promote hair regeneration by increasing the hair-inducing ability of dermal papillae (DP) cells.

The general objective of this study is to conduct a safety and feasibility study of a single injection of autologous adipose-derived SVF cells for the treatment of alopecia.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, non-blinded, interventional, consecutive series, single site study to determine initial safety and feasibility of a single injection of autologous adipose-derived SVF cells for the treatment of alopecia.

Up to 8 subjects who have been diagnosed with androgenetic alopecia will be asked to participate. Before the procedure the density (number of hairs per square centimeter) and thickness (mm) of the hair will be measured and compared to the same measurements after the procedure. All adverse events will be recorded and evaluated for severity.

Subjects will be asked to come into the office on the following days: pre-procedure visit, 24 hours post procedure visit, 6 weeks post procedure visit, 3 months post procedure visit and 6 months post procedure visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be in good health (ASA Class I-II) with a BMI < 35.
* Must have at least a 2cm x 2cm spot on the scalp which shows evidence of alopecia without scarring or traumatic injury
* Able and willing to make the required study visits.
* Able and willing to give consent and follow study instructions.
* Must speak, read and understand English

Exclusion Criteria:

* History of bleeding disorders, anticoagulation therapy that cannot be stopped 14 days prior to injection
* Allergic to lidocaine, epinephrine, Vancomycin, cephalexins, cephalosporins, penicillins, chlorhexidine gluconate, or tattoo ink
* Individuals with a propensity for keloids
* Individuals with diminished decision-making capacity will not be included in this research study.
* Current use of anti-inflammatory or anticoagulation medications that affect bleeding or are for bleeding disorders. These include: Plavix, Warfarin (Coumadin, Jantoven, Marfarin).
* Use of concomitant treatments to improve hair growth, including topical medications, oral medications, meso-therapy, non-ablative fractional laser treatment, low-level laser therapy, interfollicular PRP injection and hair transplantation within the preceding 6 months.
* Smoking and other tobacco use.
* Pregnancy or lactating period for females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 6 months
  Adverse events will be recorded and evaluated.

SECONDARY OUTCOMES:
Growth of new hair from baseline to 6 weeks, 3 months and 6 months | Changes from baseline to 6 weeks, 3 months and 6 months
  Hair density (number of hairs per square centimeter) will be measured before treatment and compared to the same measurements after treatment.
Change in hair thickness from baseline to 6 weeks, 3 months and 6 months | Changes from baseline to 6 weeks, 3 months and 6 months
  Hair thickness (mm) will be measured before treatment and compared to the same measurements after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Katz, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided